CLINICAL TRIAL: NCT00632684
Title: Adaptive Intervention for At-risk Family Caregivers
Brief Title: Effectiveness of an Adaptive Treatment Model for At-risk Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Steven H. Zarit, Penn State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH073559 (NIH); R34MH073559 (NIH); DATR A4-GPS
Record Dates: First submitted 2008-03-07; First posted 2008-03-11 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2009-04

CONDITIONS: Stress
Keywords: Family Caregiving; Dementia
MeSH Terms: conditions — Dementia | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants in Phase 1 will undergo four interviews, including a single treatment planning session.
  Interventions: Behavioral: Interviews with a single treatment planning session
- 2 (Experimental): Participants in Phase 2 will receive the adaptive treatment model.
  Interventions: Behavioral: Adaptive treatment model

INTERVENTIONS:
Behavioral: Interviews with a single treatment planning session — Participants in Phase 1 will attend four 90-minute interviews over 4 months. During interviews, participants will be asked about their experiences caring for their relatives, physical and emotional well-being, and ideas on helpful types of assistance. Participants will also receive information about programs and services that may help them carry out caregiving activities.
  Arms: 1
Behavioral: Adaptive treatment model — The adaptive treatment model will include up to ten 60- to 75-minute planning sessions. The sessions will focus on psychosocial issues and will be tailored to participants' specific risk factors.
  Arms: 2

SUMMARY:
This study will develop and evaluate the effectiveness of an adaptive treatment model for reducing the stress of, and burden on, family members caring for a person with dementia.

DETAILED DESCRIPTION:
Caring for a person with dementia can be a highly stressful experience associated with a variety of negative outcomes. Family caregivers are more likely than noncaregivers to experience symptoms of depression and anxiety, feelings of anger, and health problems. Although there are multiple treatment models to address the adverse mental and physical health outcomes associated with caregiving, most do not account for the specific risk and protective factor differences among caregivers of people with dementia. Such models provide the same treatment to all participants and have demonstrated only limited success in this high-risk caregiver population. An adaptive treatment model based on the Stress Process Model of caregiving, which emphasizes that there are multiple factors that affect stress, social support, and mental health, may better meet the needs of family caregivers. This study will first develop an adaptive treatment model, based on the Stress Process Model, for family caregivers of a person suffering from dementia. The study will then evaluate the effectiveness of each component of the adaptive treatment model in improving negative outcomes in the family caregivers.

This study will be conducted in two phases. Phase 1 will be used to develop an adaptive treatment model and risk report from which tailored treatment will be prescribed to participants in Phase 2. Participants in Phase 1 will attend four 90-minute interviews over 4 months. The first three interviews will be held in the first 3 to 4 weeks of the study and the last will be about 3 months later. In the first interview, participants will be asked about their experiences caring for their relatives, physical and emotional well-being, and ideas on helpful types of assistance. In the second and third interviews, participants will discuss their caregiving situations in more detail and will receive information about programs and services that may help them carry out caregiving activities. During the final interview, participants will again be asked about their experiences caring for their relatives.

Phase 2 of the study will test the adaptive treatment model developed in Phase 1. Participants in Phase 2 will attend an initial and final interview and up to 10 planning sessions. Each interview or planning session will last 60 to 75 minutes and will be tailored to the risks of each individual caregiver. During planning sessions, participants will discuss their caregiving situations in more detail, learn strategies to deal with stress, and receive information about programs and services that may help in carrying out caregiving activities. The strategies that participants will learn may include the following: new skills for communicating with the person receiving care, reflecting upon ways to reduce the impact of the changes that caregiving has had on their lives, learning more effective ways of communicating their own needs to other family members and friends, and identifying which types of services might be useful in caring for the person with dementia. The Phase 2 interviews will be the same as the initial and final interviews of Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a person suffering from any type of dementia and living in the community

Exclusion Criteria:

* Primary caregiver of person with late- or end-of-life stage dementia
* Primary caregiver of person with dementia who lives in skilled nursing care environment
* Primary caregiver is under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Role overload | Measured immediately after treatment

SECONDARY OUTCOMES:
Nine-Item Depression Scale of the Patient Health Questionnaire (PHQ-9) | Measured immediately after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Zarit, PhD, Principal Investigator — Penn State University; Carol J. Whitlatch, PhD, Principal Investigator — Benjamin Rose Institute
Locations (1):
- Benjamin Rose Institute, Cleveland, Ohio, United States